CLINICAL TRIAL: NCT03781908
Title: Management Of Malignant Pleural Effusion With Indwelling Pleural Catheter Versus Silver Nitrate Pleurodesis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Essmat Hussien, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: silver nitrate pleurodesis
Record Dates: First submitted 2018-11-11; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Silver Nitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Nitrate Pleurodesis (Experimental): Patients will receive 0.5% silver nitrate diluted in 50 ml distilled water with 10 ml of local anaesthetic lidocaine 1%
  Interventions: Drug: Silver Nitrate
- Indwelling Pleural Catheter (Active Comparator): Catheters will be inserted in an outpatient setting under local anaesthesia.The typical drainage schedule is every other day using disposable plastic bottles (550 mL to 1 L)
  Interventions: Device: Indwelling Pleural Catheter

INTERVENTIONS:
Drug: Silver Nitrate — First, pleural fluid drainage will be done after administration of 5 cc of local anesthetic lidocain1% either by insertion of chest tube (26F or 28F ) or by using ultrasonography. Pleural fluid drainage will be terminated when the patient want to cough to make sure that the pleural cavity is empty, then the sclerosant material will be injected, patients will receive 0.5% silver nitrate diluted in 50 ml distilled water with 10 ml of local anaesthetic lidocaine 1%.
  Arms: Silver Nitrate Pleurodesis
Device: Indwelling Pleural Catheter — First , insert the wire into the pleural effusion at approximately the anterior axillary line. A 1-2 cm incision is made over the wire. A chest wall tunnel (5-8 cm in length) is created with a counter incision. The catheter is pulled through the tunnel and out next to the wire. After dilation of the wire tract with a Teflon "peel-away" sheath, the indwelling catheter is inserted into the chest. The counter incision is closed primarily, and the catheter is secured to the skin medially with a suture.
  Arms: Indwelling Pleural Catheter

SUMMARY:
The primary goal of this study is to compare well-defined pleural effusion management success outcomes in patients with malignant or paramalignant pleural effusions who were treated with Indwelling pleural catheter insertion compared with those treated with siver nitrate pleurodesis. It is also to demonstrate the effectiveness of silver nitrate pleurodesis. It is also important to evaluate frequent adverse events of silver nitrate pleurodesis in patients with malignant pleural effusion

DETAILED DESCRIPTION:
Dyspnea is present in 50% of patients with malignant pleural effusion and quality of life is significantly impaired.

Chemical pleurodesis using various sclerosing agents is accepted as a palliative therapy for patients with recurrent, symptomatic, and malignant pleural effusions.

Silver nitrate solution (SNS) is a valid sclerosing agent that induce a caustic injury to the mesothelium that results in an effective pleurodesis.

However, various clinical parameters and biochemical factors affect the success of pleurodesis in symptomatic patients with MPE: symptoms and performance status of the patient, daily fluid drainage, primary tumour, and mainly lung reexpansion following pleural fluid evacuation.

The pleural injectate consists of 50 mL 0.5% SNS with 10mL of lidocaine (25mg/5mL).

An alternative treatment is intermittent or continuous drainage of the pleural fluid with a chronic indwelling pleural catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral symptomatic recurrent malignant pleural effusion patients who fulfill the criteria for pleurodesis (i.e. positive pleural biopsy or cytology for malignancy, a Karnofsky index score of more than 60 and life expectancy of more than one year).
2. Rapidly accumulated undiagnosed pleural effusion .
3. Age : 30-75 years old.

Exclusion Criteria:

1. Transudative pleural effusion.
2. Exudative pleural effusion due to causes other than malignancy ( i.e. parapnuemonic , post-tuberculous pleural effusion )
3. Presence of hemorrhagic diathesis ( prothrombin time <50% and platelet count <80,000/mm 3 )
4. Active pleural or systemic infection.
5. Neoplastic infiltration of the skin at the site of pleural catheter insertion.
6. Malignant pleural effusion with trapped lung or loculated pleural effusion.
7. Previous lobectomy or pneumonectomy on the affected side.
8. Karnofsky index score> 50.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of silver nitrate pleurodesis | One week
  patients will be submitted to serial chest x-ray and evaluation of pleural fluid accumulation by chest ultrasound .
Success rate of silver nitrate pleurodesis | One month
  Pleural fluid re-accumulation will be evaluated by chest x-ray and chest ultrasound.

SECONDARY OUTCOMES:
Chest pain: VAS | One week
  Chest pain will be evaluated by visual analog scale which varies from (0-10) in which grade 0 indicates no hurt and grade 10 which hurts worst
Dyspnea | One week
  Dyspnea will be evaluated through the mMRC dyspnea scale ( modified medical research council dyspnea scale) which varies from ( 0-4) in which grade 0 indicates dyspnea with sternous exercise and grade 4 which indicates dyspnea with dressing or undressing

REFERENCES:
- [Background] Kalomenidis I. Beyond talc pleurodesis: do we really need new methods? Respirology. 2011 Oct;16(7):1020-2. doi: 10.1111/j.1440-1843.2011.02023.x. No abstract available. PMID 21790880
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691
- [Background] Tremblay A, Stather DR, Kelly MM. Effect of repeated administration of low-dose silver nitrate for pleurodesis in a rabbit model. Respirology. 2011 Oct;16(7):1070-5. doi: 10.1111/j.1440-1843.2011.02007.x. PMID 21651643
- [Background] Shaw PH, Agarwal R. WITHDRAWN: Pleurodesis for malignant pleural effusions. Cochrane Database Syst Rev. 2013 Nov 20;2013(11):CD002916. doi: 10.1002/14651858.CD002916.pub3. PMID 24259053
- [Background] Arber A, Clackson C, Dargan S. Malignant pleural effusion in the palliative care setting. Int J Palliat Nurs. 2013 Jul;19(7):320, 322-5. PMID 24273808
- [Background] Suarez PM, Gilart JL. Pleurodesis in the treatment of pneumothorax and pleural effusion. Monaldi Arch Chest Dis. 2013 Jun;79(2):81-6. doi: 10.4081/monaldi.2013.96. PMID 24354096
- [Background] Schneider T, Reimer P, Storz K, Klopp M, Pfannschmidt J, Dienemann H, Hoffmann H. Recurrent pleural effusion: who benefits from a tunneled pleural catheter? Thorac Cardiovasc Surg. 2009 Feb;57(1):42-6. doi: 10.1055/s-2008-1039109. Epub 2009 Jan 23. PMID 19169996
- [Background] Ferlay JSH, Bray F, Forman D, Mathers C, Parkin DM, eds. Cancer incidence and mortality worldwide [webpage]. World Health Organization, International Agency for Research on Cancer; 2008. v1.2. CancerBase No. 10. http://globocan.iarc.fr. Accessed November 11, 2011.
- [Background] Light RW, Vargas FS. Pleural sclerosis for the treatment of pneumothorax and pleural effusion. Lung. 1997;175(4):213-23. doi: 10.1007/pl00007568. PMID 9195549